CLINICAL TRIAL: NCT03100955
Title: A Study of Standard Treatment +/- Apatinib in Extensive Stage Small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qingdao University (Other)
Responsible Party: Principal Investigator, medley nie, Secretary of clinical trials, Qingdao University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QU20170327
Record Dates: First submitted 2017-03-26; First posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Progression Free Survival
MeSH Terms: interventions — PE regimen; Cisplatin; Etoposide; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EP chemotherapy (Active Comparator): Standard treatment or active comparator group contains a platinum drug and a topoisomerase inhibitor. Platinum drug=cisplatin 75 mg/m2 iv on day 1; topoisomerase inhibitor=etoposide 120 mg/m2 iv day 1-3, 3 weeks a cycle, total numbers of cycles 6.Used drugs=cisplatinum and etoposide.
  Interventions: Drug: cisplatin, etoposide
- EP chemotherapy plus apatinib (Experimental): Apatinib treatment or experimental group contains standard chemotherapy and apatinib, a VEGF tyrosine kinase inhibitor. It contains a platinum drug, a topoisomerase inhibitor and a VEGF-TKI. Platinum drug=cisplatin 75 mg/m2 iv on day 1; topoisomerase inhibitor=etoposide 120 mg/m2 iv day 1-3, 3 weeks a cycle, total numbers of cycles 6.Used drugs=cisplatinum and etoposide. Numbers of cycles 6. In addition to this, subjects will receive VEGF-TKI=apatinib, 500 mg, oral daily after chemotherapy, until disease progression or death or un-tolerated toxicites. Used drugs=cisplatinum and etoposide and apatinib.
  Interventions: Drug: cisplatin, etoposide, apatinib

INTERVENTIONS:
Drug: cisplatin, etoposide — The recommended regimen is cisplatin plus etoposide. cisplatin 75 mg/m2 iv on day 1, etoposide 120 mg/m2 iv on day 1-3, 3 weeks a cycle, total for 6 cycles is allowed.
  Arms: EP chemotherapy
Drug: cisplatin, etoposide, apatinib — Standard chemotherapy treatment for patients with small cell lung cancer. Chemotherapy regimen contains a platinum drug and a topoisomerase inhibitor. Platinum drug=cisplatin 75 mg/m2 iv on day 1; topoisomerase inhibitor=etoposide 120 mg/m2 iv day 1-3, 3 weeks a cycle, total numbers of cycles 6.Used drugs=cisplatin and etoposide. Numbers of cycles 6. In addition to this, subjects will receive VEGF-TKI apatinib oral daily after chemotherapy treatment. Apatinib 500mg oral, once a day, until disease progression or death or un-tolerated toxicites.
  Arms: EP chemotherapy plus apatinib

SUMMARY:
To establish the progression free survival in patients with extensive stage small cell lung cancer treated with cisplatin and etoposide plus or not apatinib

DETAILED DESCRIPTION:
Assess progression free survival, overall survival and toxicity of standard EP regimen combined or not with VEGF tyrosine kinase inhibitor-apatinib. Response measured by RECIST response criteria. Toxicity via physical exam, adverse event review, assessing signs and symptoms, quality of life assessment and blood testing.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically verified SCLC, extensive stages
2. WHO performance status 0, 1, 2
3. Age 18 years or older
4. Treatment naive
5. Anticipated survival more than 3 months
6. HB >90g/L, ANC>1.5 x 109/L, Platelets >80 x109 /L
7. No prognancy
8. Signed informed consent

Exclusion Criteria:

1. Limited stage disease
2. Metastastic meningitis, spinal compression, Tumor to main vesicular less than 5mm
3. Uncontrolled hypertension
4. Uncontrolled heart failure
5. Coagulation problem
6. Surgery, trauma, uncontrolled ulcer in 4 weeks.
7. Required by physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 24 months
  from the date of randomization to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Zhuang Yu, MD, Ph. D, Study Chair — The Affiliated Hospital of Qingdao University
Locations (1):
- Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No